CLINICAL TRIAL: NCT05186922
Title: A Randomized, Double Blind, Placebo-Controlled, Multiple Dose Escalation, Phase 2 Study to Evaluate the Safety, Tolerance, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Preliminary Efficacy of CM326 in Patients With Moderate-severe Atopic Dermatitis Subjects
Brief Title: The Study of CM326 in Patients With Moderate-to-severe Atopic Dermatitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM326AD001
Record Dates: First submitted 2021-12-13; First posted 2022-01-11 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Moderate-to-severe Atopic Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CM326 55 mg, once every two weeks (Q2W) (Experimental): 55mg for 6 doses, every 2 weeks, subcutaneous (SC)
  Interventions: Biological: CM326
- CM326 110 mg, once every two weeks (Q2W) (Experimental): 110mg for 6 doses, every 2 weeks, subcutaneous (SC)
  Interventions: Biological: CM326
- CM326 110 mg, once every four weeks (Q4W) (Experimental): 110mg for 3 doses, every 4 weeks, subcutaneous (SC)
  Interventions: Biological: CM326
- CM326 220 mg, once every two weeks (Q2W) (Experimental): 220mg for 6 doses, every 2 weeks, subcutaneous (SC)
  Interventions: Biological: CM326
- CM326 220 mg, once every four weeks (Q4W) (Experimental): 220mg for 3 doses, every 4 weeks, subcutaneous (SC)
  Interventions: Biological: CM326
- Placebo (Placebo Comparator): Placebo for 6 doses, every 2 weeks, subcutaneous (SC) and placebo for 3 doses, every 4 weeks, subcutaneous (SC)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CM326 — CM326 injection
  Arms: CM326 110 mg, once every four weeks (Q4W); CM326 110 mg, once every two weeks (Q2W); CM326 220 mg, once every four weeks (Q4W); CM326 220 mg, once every two weeks (Q2W); CM326 55 mg, once every two weeks (Q2W)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled multiple dose escalation study to evaluate the safety, tolerance, PK, PD, immunogenicity and preliminary efficacy of CM326 in moderate-severe AD subjects.

DETAILED DESCRIPTION:
The study consists of 3 periods, a up-to-4-week Screening Period, a 12-week randomized Treatment Period and a 12-week Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed Atopic Dermatitis (AD) at least 12 months before the screening
* Eczema Area and Severity Index (EASI) score ≥16 at screening and baseline
* Investigator's Global Assessment (IGA) score ≥3 at screening and baseline
* Body Surface Area (BSA) of involvement of atopic dermatitis ≥10% at screening and baseline
* The weekly mean score of daily peaks in pruritus NRS at baseline ≥4
* Provide signed informed consent

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Presence of other concomitant and poorly controlled serious diseases or recurrent chronic diseases, including but not limited to active infections, cardiovascular and cerebrovascular diseases, pulmonary tuberculosis or other pathogen infections, diabetes mellitus, autoimmune diseases, human immunodeficiency virus (HIV) infection, active hepatitis B, hepatitis C or parasitosis, neoplasm malignant, etc.
* Patients with severe hepatic or renal impairment, characterized by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > 2 times of upper limit of normal (ULN), total bilirubin >1.5 times of upper limit of normal (ULN) or serum creatinine level > upper limit of normal (ULN).
* Womens who are pregnant or breastfeeding, or who plan to become pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AE) | Up to week 24
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter: Time to reach peak concentration (Tmax) | Up to Week 24
  Time to reach peak concentration (Tmax)
Pharmacokinetics (PK) parameter : Peak Plasma concentration (Cmax) | Up to Week 24
  Peak Plasma concentration (Cmax)
Pharmacokinetics (PK) parameter : Area under the plasma concentration-time curve (AUC) | Up to Week 24
  Area under the plasma concentration-time curve (AUC)
Pharmacokinetics (PK) parameter : Clearance rate (CL/F) | Up to Week 24
  Clearance rate (CL/F)
Pharmacokinetics (PK) parameter : Elimination half life (T1/2z) | Up to Week 24
  Elimination half life (T1/2z)
Pharmacodynamics (PD): Changes from baseline in serum thymus activation regulation chemokine (TARC) concentration after CM326 administration | Up to Week 24
  Changes from baseline in serum thymus activation regulation chemokine (TARC) concentration after CM326 administration
Pharmacodynamics (PD): Changes from baseline in eosinophil count after CM326 administration | Up to Week 24
  Changes from baseline in eosinophil count after CM326 administration
Pharmacodynamics (PD): Changes from baseline in serum total immunoglobulin E (IgE) concentration after CM326 administration | Up to Week 24
  Changes from baseline in serum total immunoglobulin E (IgE) concentration after CM326 administration
Pharmacodynamics (PD): Changes from baseline in plasma interleukin-5 (IL-5) concentration after CM326 administration | Up to Week 24
  Changes from baseline in plasma interleukin-5 (IL-5) concentration after CM326 administration
Pharmacodynamics (PD): Changes from baseline in plasma interleukin-13 (IL-13) concentration after CM326 administration | Up to Week 24
  Changes from baseline in plasma interleukin-13 (IL-13) concentration after CM326 administration
Pharmacodynamics (PD): Changes from baseline in serum periostin concentration after CM326 administration | Up to Week 24
  Changes from baseline in serum periostin concentration after CM326 administration
Immunogenicity: anti-drug antibody (ADA) and neutralizing antibody (Nab) | Up to Week 24
  Detection of anti-drug antibody (ADA) and neutralizing antibody (Nab)
Proportion of patients with Investigator's Global Assessment (IGA) score = 0-1 at each visit | Up to Week 24
  IGA is a 6-point scale ranging from 0 (clear) to 5 (very severe)
Proportion of patients with IGA reduction from baseline of ≥2 points at each visit | Up to Week 24
  IGA is a 6-point scale ranging from 0 (clear) to 5 (very severe)
Proportion of patients with Eczema Area and Severity Index (EASI)-50 (≥50 percent reduction in EASI scores from baseline) at each visit | Up to Week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Eczema Area and Severity Index (EASI)-75 (≥75 percent reduction in EASI scores from baseline) at each visit | Up to Week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with Eczema Area and Severity Index (EASI)-90 (≥90 percent reduction in EASI scores from baseline) at each visit | Up to Week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Change from baseline in Eczema Area and Severity Index (EASI) score at each visit | Up to Week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 to 72 points, with the higher scores reflecting the worse severity of AD
Proportion of patients with reduction of Pruritus Numerical Rating Scale (NRS) of ≥3 and ≥4 points from baseline | Up to Week 24
  The range of NRS is from 0 (no itch)-10 (worst imaginable itch)
Percent change from baseline in Numerical Rating Scale (NRS) | Up to Week 24
  The range of NRS is from 0 (no itch)-10 (worst imaginable itch)
Body surface area (BSA) of involvement of atopic dermatitis | Up to Week 24
  Change from baseline in percent of BSA
Changes from baseline in Dermatology Life Quality Index (DLQI) at each visit | Up to Week 24
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's hospital, Beijing, Beijing Municipality, China